CLINICAL TRIAL: NCT05000944
Title: Impact of Breakfast Consumption Timing on Postprandial Glycaemia and Insulinaemia in Adolescent Girls Who Habitually Skip Breakfast
Brief Title: Is Mid-morning Breakfast as Healthy as Early-morning Breakfast for Blood Sugar Control in Adolescent Girls?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Sahar Afeef, PhD student, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 3129
Record Dates: First submitted 2021-07-30; First posted 2021-08-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Postprandial Hyperglycemia
Keywords: Breakfast; Meal Time; Blood Glucose; Blood Insulin; Adolescents
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: same participants will complete three breakfast conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- breakfast omission (BO) (Experimental): No breakfast will be provided until the lunch time at ~12:30. Blood samples will be taken at fasting state and postprandially at different intervals after breakfast and lunch for the measurement of glucose and insulin concentrations.
  Interventions: Other: breakfast omission (BO)
- early-morning breakfast consumption (EM-BC) (Experimental): A standardised, carbohydrate-rich, low glycaemic index (GI) breakfast will be provided at ~08:30 for EM-BC. Blood samples will be taken at fasting state and postprandially at different intervals after breakfast and lunch for the measurement of glucose and insulin concentrations.
  Interventions: Other: early-morning breakfast consumption (EM-BC)
- mid-morning breakfast consumption (MM-BC). (Experimental): A standardised, carbohydrate-rich, low glycaemic index (GI) breakfast will be provided at ~10:30 for MM-BC (i.e., two hours after EM-BC). Blood samples will be taken at fasting state and postprandially at different intervals after breakfast and lunch for the measurement of glucose and insulin concentrations.
  Interventions: Other: mid-morning breakfast consumption (MM-BC)

INTERVENTIONS:
Other: breakfast omission (BO) — this group will not be provided with a breakfast until lunch time (at 12:30).
  Other Names: skipping breakfast
  Arms: breakfast omission (BO)
Other: early-morning breakfast consumption (EM-BC) — this group will be provided with an early morning breakfast (at 08:30).
  Other Names: early breakfast
  Arms: early-morning breakfast consumption (EM-BC)
Other: mid-morning breakfast consumption (MM-BC) — this group will be provided with a mid (late) morning breakfast (at 10:30).
  Other Names: late breakfast
  Arms: mid-morning breakfast consumption (MM-BC).

SUMMARY:
Repeated, elevated levels of glucose (sugar) within the blood after eating can lead to type 2 diabetes. In adults, eating breakfast lowers blood glucose responses to subsequent meals when compared with skipping breakfast. Yet, adolescent girls may respond differently due to differences in how their bodies use energy. This is important because around 80% of the United Kingdom (UK) adolescent girls skip breakfast. As common reasons for skipping breakfast in adolescent girls are 'lack of time' and 'not hungry' in the morning, eating breakfast during the mid-morning may be an attractive option for them. This project will be the first to compare the impact of eating breakfast in the early morning and mid-morning with skipping breakfast on subsequent blood glucose levels in adolescent girls who usually skip breakfast. The findings will inform recommendations tailored to an 'at risk' and under-researched population for type 2 diabetes prevention, which is more effective than a cure.

DETAILED DESCRIPTION:
Dietary manipulations that can moderate postprandial glycaemia and insulinaemia are at the cornerstone of type 2 diabetes (T2D) prevention. Indeed, repeated glycaemic excursions cause oxidative stress, inflammation, and atherosclerosis, increasing T2D risk. Adolescence is a critical time to promote dietary behaviours that can be sustained across the lifespan. Among the dietary factors influencing postprandial glycaemia, the decline in breakfast consumption during adolescence in girls is of concern, with only ~20% of UK adolescent girls consuming breakfast daily. Cross-sectional and prospective observational studies show that infrequent breakfast consumption is associated with T2D risk markers (e.g., glucose, insulin) in adolescents and T2D manifestation in adults. Randomised controlled trials in adults suggest that improvements in glycaemic control and insulin sensitivity may be key to explaining the reduced T2D risk when contrasting breakfast consumption with breakfast omission. Acutely, breakfast omission exaggerates glycaemic and insulinaemic responses to subsequent meals when compared to breakfast consumption, which has been termed the 'second-meal effect'. Thus, two moderate glycaemic responses (with breakfast and lunch) would be potentially better for reducing T2D risk than one very large glycaemic excursion (after lunch). Yet, findings based on adults may not apply to the distinct hormonal and metabolic profiles of adolescent girls. Specifically, it is proposed that the 'second-meal effect' occurs due to increased glucose conversion into muscle glycogen in adults. Such responses may differ in adolescents due to their higher reliance on exogenous glucose and fat as fuels with a lower reliance on endogenous glucose and reduced capacity for muscle glycogen storage, in addition to the 32% reduction in insulin sensitivity occurring from pre- to mid-puberty. Unfortunately, current knowledge on breakfast and glycaemia in adolescents relies entirely on a few novel studies that have pooled data from 13 to 20 year olds with little consideration of pubertal status and sex. Hence, the glycaemic responses to breakfast manipulation in adolescent girls are not still well understood. Common barriers to consuming breakfast among adolescent girls include not being hungry and a lack of time in the morning. As such, the option to consume breakfast later in the morning may be an attractive alternative for this population. In terms of timing, definitions have proposed that breakfast is consumed within 2-3 hours of waking, typically no later than 10:00. Yet, inconsistent definitions have been employed across the literature, mainly because evidence to inform a health-based (e.g., focused on glycaemic improvements) breakfast timing 'cut-off' is lacking. Thus, the unique contribution of this proposal is the use of an experimental cross-over design to directly contrast the effects of consuming an early-morning versus mid-morning standardised breakfast with breakfast omission on postprandial glycaemia and insulinaemia in adolescent girls classified as habitual breakfast skippers. By focusing on adolescent girls, breakfast timing and postprandial glycaemia, this proposal is unique, topical and has potential impact for T2D prevention.

Recruitment:

Girls will be recruited from local schools after gaining parental informed consent and child assent. These schools have expressed an interest in facilitating recruitment for the proposed research by providing a platform to invite girls to participate and permission for time off school to complete the measures. The participants will be invited to attend an assembly at their school and those that wish to discuss their participation with a parent/primary caregiver will take an information pack home that includes written details of the study. On return of a contact form, students and their primary caregiver will be asked to complete the consent, assent and pre-participation health screen questionnaire, before registration on the study.

Experimental design:

This study will employ a cross-over design. Participants will complete three conditions assigned according to the Latin square method: breakfast omission (BO), early-morning breakfast consumption (EM-BC) and mid-morning breakfast consumption (MM-BC). The conditions will be conducted ~7 days apart in girls who have not started their menses or in the early-follicular phase (~28 days apart) in girls with regular menses to minimise the potential confounding influence of menstrual cycle phase. In the 48 hours before the conditions, dietary intakes, bed time and wake/out of bed times will be replicated, and vigorous physical activity will be minimised (as confirmed via accelerometry).

After an overnight fast, resting metabolic rate (RMR) and substrate oxidation will be estimated via expired air analysis, and a capillary blood sample for the measurement of plasma glucose and insulin will be taken (~08:15 to 08:30). These measures will be collected at regular intervals, with a standardised lunch consumed at 4 h (~12:30) and followed by a 2-h lunch postprandial period. The standardised breakfast will be provided immediately after fasting measures at ~08:30 for EM-BC and 2 hours later at ~10:30 for MM-BC. Participants will remain sedentary throughout. Water intake will be replicated between the conditions.

Test meals:

A carbohydrate-rich, low glycaemic index (GI) breakfast providing ~70% carbohydrate, ~17% fat and ~13% protein will be used. The breakfast will be provided in quantities containing 0.04 g carbohydrate per kcal of individualised daily RMR. The standardised lunch providing 0.05 g of carbohydrate per kcal of daily RMR will be based on high GI carbohydrate. Meal consumption time will be limited to 15 minutes and replicated between the conditions.

Data and statistical analyses:

Pre-lunch (4 hours) and post-lunch (2 hours) incremental (iAUC) and total (tAUC) area under the curve will be calculated using the trapezium rule for the primary outcomes, plasma glucose and insulin. and the secondary outcomes, resting energy expenditure and substrate oxidation rates. In addition, peak plasma glucose concentration after lunch will be determined.

Linear mixed models will be used to compare all outcome variables between the conditions. Models will include fixed effects for condition (and time for the condition by time analyses) and a random intercept for participants, and will be adjusted for the order effect. The Holm-Bonferroni correction for multiple comparisons will be applied. Normality will be checked using Shapiro Wilk tests. Statistical significance will be accepted at p≤0.05. Cohen's effect sizes will be used to gauge the magnitude of differences.

Sample size estimation:

Based on 80% power at an alpha level of p=0.05, it is estimated that 21 breakfast skipping adolescent girls are required to detect a meaningful between-condition difference (Cohen's f=0.36) in post-lunch plasma glucose area under the curve. Recruitment will target 27 participants across the two study sites to account for an expected 20% attrition rate.

ELIGIBILITY:
Inclusion criteria:

* Girls classified habitual breakfast skippers (using a proposed definition of 'breakfast', the girls will be classified as habitual breakfast skipper if they consume breakfast 0-3 times per week)
* no health issues that could be affected by study participation (e.g., food allergies)
* no extreme dislikes of the test meals.

Exclusion criteria:

* Medical conditions or current medication that affects glucose metabolism
* Food allergies that would prevent consumption of prescribed meals

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Incremental and total area under the curve for glucose | 4 hours before lunch and 2 hours after lunch
  Blood samples will be collected at fasting and at different intervals before and after lunch meal. [Glucose] will be used to calculate 4 hours pre-lunch and 2 hours post-lunch incremental (IAUC) and total (TAUC) area under the curve using the trapezium rule.
Incremental and total area under the curve for insulin | 4 hours before lunch and 2 hours after lunch
  Blood samples will be collected at fasting and at different intervals before and after lunch meal. [Insulin] will be used to calculate 4 hours pre-lunch and 2 hours post-lunch incremental (IAUC) and total (TAUC) area under the curve using the trapezium rule.
Post-lunch peak plasma glucose concentration | 2 hours after lunch
  The highest plasma glucose concentration value during 2 hours after lunch will be determined and compared between breakfast conditions

SECONDARY OUTCOMES:
Substrate oxidation rates | 4 hours before lunch and 2 hours after lunch
  Expired gas will be collected to calculate the rates of substrate oxidation
Resting energy expenditure | 4 hours before lunch and 2 hours after lunch
  Expired gas will be collected to calculate the resting energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Keith Tolfrey, Dr, Principal Investigator — Loughborough University; Sahar Afeef, MSc, Principal Investigator — Loughborough University; Julia Zakrzewski-Fruer, Dr, Principal Investigator — University of Bedfordshire; Laura Barrett, Dr, Principal Investigator — Loughborough University
Locations (1):
- Local schools, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balk EM, Earley A, Raman G, Avendano EA, Pittas AG, Remington PL. Combined Diet and Physical Activity Promotion Programs to Prevent Type 2 Diabetes Among Persons at Increased Risk: A Systematic Review for the Community Preventive Services Task Force. Ann Intern Med. 2015 Sep 15;163(6):437-51. doi: 10.7326/M15-0452. PMID 26167912
- [Background] Dyson PA, Kelly T, Deakin T, Duncan A, Frost G, Harrison Z, Khatri D, Kunka D, McArdle P, Mellor D, Oliver L, Worth J; Diabetes UK Nutrition Working Group. Diabetes UK evidence-based nutrition guidelines for the prevention and management of diabetes. Diabet Med. 2011 Nov;28(11):1282-8. doi: 10.1111/j.1464-5491.2011.03371.x. PMID 21699560
- [Background] Heine RJ, Balkau B, Ceriello A, Del Prato S, Horton ES, Taskinen MR. What does postprandial hyperglycaemia mean? Diabet Med. 2004 Mar;21(3):208-13. doi: 10.1111/j.1464-5491.2004.01149.x. PMID 15008828
- [Background] Todd AS, Street SJ, Ziviani J, Byrne NM, Hills AP. Overweight and obese adolescent girls: the importance of promoting sensible eating and activity behaviors from the start of the adolescent period. Int J Environ Res Public Health. 2015 Feb 17;12(2):2306-29. doi: 10.3390/ijerph120202306. PMID 25690003
- [Background] Corder K, van Sluijs EM, Ridgway CL, Steele RM, Prynne CJ, Stephen AM, Bamber DJ, Dunn VJ, Goodyer IM, Ekelund U. Breakfast consumption and physical activity in adolescents: daily associations and hourly patterns. Am J Clin Nutr. 2014 Feb;99(2):361-8. doi: 10.3945/ajcn.111.027607. Epub 2013 Nov 27. PMID 24284440
- [Background] Timlin MT, Pereira MA, Story M, Neumark-Sztainer D. Breakfast eating and weight change in a 5-year prospective analysis of adolescents: Project EAT (Eating Among Teens). Pediatrics. 2008 Mar;121(3):e638-45. doi: 10.1542/peds.2007-1035. PMID 18310183
- [Background] Ballon A, Neuenschwander M, Schlesinger S. Breakfast Skipping Is Associated with Increased Risk of Type 2 Diabetes among Adults: A Systematic Review and Meta-Analysis of Prospective Cohort Studies. J Nutr. 2019 Jan 1;149(1):106-113. doi: 10.1093/jn/nxy194. PMID 30418612
- [Background] Hallstrom L, Labayen I, Ruiz JR, Patterson E, Vereecken CA, Breidenassel C, Gottrand F, Huybrechts I, Manios Y, Mistura L, Widhalm K, Kondaki K, Moreno LA, Sjostrom M; HELENA Study Group. Breakfast consumption and CVD risk factors in European adolescents: the HELENA (Healthy Lifestyle in Europe by Nutrition in Adolescence) Study. Public Health Nutr. 2013 Jul;16(7):1296-305. doi: 10.1017/S1368980012000973. Epub 2012 Apr 12. PMID 22494882
- [Background] Smith KJ, Gall SL, McNaughton SA, Blizzard L, Dwyer T, Venn AJ. Skipping breakfast: longitudinal associations with cardiometabolic risk factors in the Childhood Determinants of Adult Health Study. Am J Clin Nutr. 2010 Dec;92(6):1316-25. doi: 10.3945/ajcn.2010.30101. Epub 2010 Oct 6. PMID 20926520
- [Background] Betts JA, Richardson JD, Chowdhury EA, Holman GD, Tsintzas K, Thompson D. The causal role of breakfast in energy balance and health: a randomized controlled trial in lean adults. Am J Clin Nutr. 2014 Aug;100(2):539-47. doi: 10.3945/ajcn.114.083402. Epub 2014 Jun 4. PMID 24898233
- [Background] Chowdhury EA, Richardson JD, Tsintzas K, Thompson D, Betts JA. Carbohydrate-rich breakfast attenuates glycaemic, insulinaemic and ghrelin response to ad libitum lunch relative to morning fasting in lean adults. Br J Nutr. 2015 Jul 14;114(1):98-107. doi: 10.1017/S0007114515001506. Epub 2015 May 25. PMID 26004166
- [Background] Chowdhury EA, Richardson JD, Holman GD, Tsintzas K, Thompson D, Betts JA. The causal role of breakfast in energy balance and health: a randomized controlled trial in obese adults. Am J Clin Nutr. 2016 Mar;103(3):747-56. doi: 10.3945/ajcn.115.122044. Epub 2016 Feb 10. PMID 26864365
- [Background] Boisseau N, Delamarche P. Metabolic and hormonal responses to exercise in children and adolescents. Sports Med. 2000 Dec;30(6):405-22. doi: 10.2165/00007256-200030060-00003. PMID 11132123
- [Background] Jovanovic A, Leverton E, Solanky B, Ravikumar B, Snaar JE, Morris PG, Taylor R. The second-meal phenomenon is associated with enhanced muscle glycogen storage in humans. Clin Sci (Lond). 2009 Jul 2;117(3):119-27. doi: 10.1042/CS20080542. PMID 19161346
- [Background] Timmons BW, Bar-Or O, Riddell MC. Oxidation rate of exogenous carbohydrate during exercise is higher in boys than in men. J Appl Physiol (1985). 2003 Jan;94(1):278-84. doi: 10.1152/japplphysiol.00140.2002. Epub 2002 Sep 13. PMID 12391100
- [Background] Timmons BW, Bar-Or O, Riddell MC. Energy substrate utilization during prolonged exercise with and without carbohydrate intake in preadolescent and adolescent girls. J Appl Physiol (1985). 2007 Sep;103(3):995-1000. doi: 10.1152/japplphysiol.00018.2007. Epub 2007 Jul 5. PMID 17615283
- [Background] Goran MI, Gower BA. Longitudinal study on pubertal insulin resistance. Diabetes. 2001 Nov;50(11):2444-50. doi: 10.2337/diabetes.50.11.2444. PMID 11679420
- [Background] Alwattar AY, Thyfault JP, Leidy HJ. The effect of breakfast type and frequency of consumption on glycemic response in overweight/obese late adolescent girls. Eur J Clin Nutr. 2015 Aug;69(8):885-90. doi: 10.1038/ejcn.2015.12. Epub 2015 Feb 25. PMID 25711955
- [Background] Bauer LB, Reynolds LJ, Douglas SM, Kearney ML, Hoertel HA, Shafer RS, Thyfault JP, Leidy HJ. A pilot study examining the effects of consuming a high-protein vs normal-protein breakfast on free-living glycemic control in overweight/obese 'breakfast skipping' adolescents. Int J Obes (Lond). 2015 Sep;39(9):1421-4. doi: 10.1038/ijo.2015.101. Epub 2015 Jun 1. PMID 26028058
- [Background] Shaw ME. Adolescent breakfast skipping: an Australian study. Adolescence. 1998 Winter;33(132):851-61. PMID 9886013
- [Background] O'Neil CE, Byrd-Bredbenner C, Hayes D, Jana L, Klinger SE, Stephenson-Martin S. The role of breakfast in health: definition and criteria for a quality breakfast. J Acad Nutr Diet. 2014 Dec;114(12 Suppl):S8-S26. doi: 10.1016/j.jand.2014.08.022. Epub 2014 Nov 24. No abstract available. PMID 25458994
- [Background] Timlin MT, Pereira MA. Breakfast frequency and quality in the etiology of adult obesity and chronic diseases. Nutr Rev. 2007 Jun;65(6 Pt 1):268-81. doi: 10.1301/nr.2007.jun.268-281. PMID 17605303
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Deleterious effects of omitting breakfast on insulin sensitivity and fasting lipid profiles in healthy lean women. Am J Clin Nutr. 2005 Feb;81(2):388-96. doi: 10.1093/ajcn.81.2.388. PMID 15699226